CLINICAL TRIAL: NCT01317875
Title: A Phase Ib, Open-label, Dose-finding Study of the JAK Inhibitor INC424 Tablets Administered Orally to Patients With Primary Myelofibrosis (PMF), Post-polycythemia Veramyelofibrosis (PPV-MF) or Post-essentialthrombocythemia-myelofibrosis (PET-MF) and Baseline Platelet Counts ≥50 x109/L and <100 x109/L (EXPAND)
Brief Title: Study of the JAK Inhibitor Ruxolitinib Administered Orally to Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera-Myelofibrosis (PPV-MF) or Post-Essential Thrombocythemia-Myelofibrosis (PET-MF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2201; 2010-023055-29 (EudraCT Number)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2011-03-14; First posted 2011-03-17 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum -1 (Experimental): Participants with baseline Platelet counts of 75-99 x10^9/L
  Interventions: Drug: Ruxolitinib
- Stratum -2 (Experimental): Participants with baseline Platelet counts of 50-74 x10^9/L
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Starting dose of ruxolitinib for cohort 1 in dose escalation phase - 5mg twice a day (BID)
  Doses will be increased a total of approximately 5mg for successive dosing cohorts based on baseline platelet count
  Other Names: INCB018424

SUMMARY:
This is a Phase IB, open-label, dose-finding study of the JAK 1 and 2 inhibitor ruxolitinib in patients with myelofibrosis (MF). The study consists of two periods: the core study period, comprising the dose escalation stage and the safety extension phase up to Week 24, then the extension study period beyond Week 24 and up to 3 years, to further characterize the safety and efficacy of ruxolitinib in this patient population. The dose escalation phase will enroll successive cohorts of patients who receive increasing doses of ruxolitinib until the maximum safe starting dose (MSSD) is determined. In the safety expansion phase, additional patients will be treated with ruxolitinib at the MSSD defined during dose escalation. The primary objective is to establish the MSSD of ruxolitinib in patients with MF and starting platelet counts < 100 x 10 ^9/L

ELIGIBILITY:
Inclusion Criteria:

* Require treatment for MF and classified at least as intermediate risk level 1 defined by the International Working Group.
* Platelet count < 100x10 ^9/L at screening or at Study Day 1.

Exclusion Criteria:

* Received platelet transfusion within 14 days prior to Screening evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (18):
- United States (3):
  - Winter Park, Florida
  - Baltimore, Maryland
  - Houston, Texas
- Vienna, Austria
- China (4):
  - Nanjing, Jiangsu
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
- France (3):
  - Angers
  - Paris
  - Pierre-Bénite
- Leipzig, Germany
- Italy (3):
  - Florence
  - Milan
  - Terni
- Rotterdam, Netherlands
- United Kingdom (2):
  - Belfast
  - London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guglielmelli P, Kiladjian JJ, Vannucchi AM, Duan M, Meng H, Pan L, He G, Verstovsek S, Boyer F, Barraco F, Niederwieser D, Pungolino E, Liberati AM, Harrison C, Roussou P, Wroclawska M, Karumanchi D, Sinclair K, Te Boekhorst PAW, Gisslinger H. Efficacy and safety of ruxolitinib in patients with myelofibrosis and low platelet count (50 x 109/L to <100 x 109/L) at baseline: the final analysis of EXPAND. Ther Adv Hematol. 2022 Sep 10;13:20406207221118429. doi: 10.1177/20406207221118429. eCollection 2022. PMID 36105914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 03-Mar-2011 to 31-Dec-2019 globally. Participants with MF and baseline PLT of 75 to < 100 × 109/L are enrolled in Stratum 1;and 50 to < 75 × 109/L are enrolled in Stratum 2.. The study has a core period (up to week 24) consisting of 2 phases (dose escalation and safety expansion) followed by an extension period (up to 3 years). Participants received increasing doses of ruxolitinib until the Maximum Safe Starting Dose (MSSD) was determined
Pre-assignment Details: A total of 69 participants enrolled in the study with 44 in Stratum 1 (cohorts 1,2,3,4,5) and 25 in Stratum 2 (Cohorts 1,2,3).
Groups:
- Stratum 1 : Cohort 1: Ruxolitinib was administered at 5 mg bid in Participants with baseline Platelet counts of 75-99x10^9/L
- Stratum 1 : Cohort 2: Ruxolitinib was administered at 5 mg q.AM / 10 mg q.PM in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 1 : Cohort 3: Ruxolitinib was administered to cohort 3 at 10 mg bid in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 1 : Cohort 4: Ruxolitinib was administered at 10 mg q.AM / 15 mg q.PM in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 1 : Cohort 5: Ruxolitinib was administered at 15 mg bid in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 2 : Cohort 1: Ruxolitinib was administered at 5 mg bid in participants with baseline Platelet counts of 50-74x10^9/L
- Stratum 2 : Cohort 2: Ruxolitinib was administered at 5 mg q.AM / 10 mg q.PM in participants with baseline Platelet counts of 50-74 x10^9/L
- Stratum 2 : Cohort 3: Ruxolitinib was administered at 10 mg bid in participants with baseline Platelet counts of 50-74 x10^9/L
- Stratum 2 : Cohort 4: Ruxolitinib was administered at 10 mg q.AM / 15 mg q.PM in participants with baseline Platelet counts of 50-74 x10^9/L
- Stratum 2 : Cohort 5: Ruxolitinib was administered at 15 mg bid in participants with baseline Platelet counts of 50-74 x10^9/L
Period: Overall Study
Arm/Group | Stratum 1 : Cohort 1 | Stratum 1 : Cohort 2 | Stratum 1 : Cohort 3 | Stratum 1 : Cohort 4 | Stratum 1 : Cohort 5 | Stratum 2 : Cohort 1 | Stratum 2 : Cohort 2 | Stratum 2 : Cohort 3 | Stratum 2 : Cohort 4 | Stratum 2 : Cohort 5
Started | 5 | 3 | 20 | 4 | 12 | 3 | 4 | 18 | 0 (No participants enrolled in Stratum 2 : Cohort 4) | 0 (No participants enrolled in Stratum 2 : Cohort 5)
Completed | 2 | 1 | 11 | 2 | 3 | 1 | 2 | 3 | 0 | 0
Not Completed | 3 | 2 | 9 | 2 | 9 | 2 | 2 | 15 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance with study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 2 | 1 | 5 | 1 | 2 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Stratum 1 : Cohort 4: Ruxolitinib was administered at 10 mg q.AM / 15 mg q.PM) in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 2 : Cohort 2: Ruxolitinib was administered at 5 mg q.AM / 10 mg q.PM) in participants with baseline Platelet counts of 50-74 x10^9/L
- Total: Total of all reporting groups
Arm/Group | Stratum 1 : Cohort 1 | Stratum 1 : Cohort 2 | Stratum 1 : Cohort 3 | Stratum 1 : Cohort 4 | Stratum 1 : Cohort 5 | Stratum 2 : Cohort 1 | Stratum 2 : Cohort 2 | Stratum 2 : Cohort 3 | Stratum 2 : Cohort 4 | Stratum 2 : Cohort 5 | Total
Number analyzed (Participants) | 5 | 3 | 20 | 4 | 12 | 3 | 4 | 18 | 0 | 0 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.00 (7.78) | 54.00 (4.00) | 63.0 (14.71) | 70.4 (8.91) | 75.8 (3.30) | 67.3 (11.06) | 72.5 (6.95) | 68.0 (11.66) |  |  | 66.4 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 12 | 2 | 4 | 2 | 3 | 7 |  |  | 36
  Male | 1 | 1 | 8 | 2 | 8 | 1 | 1 | 11 |  |  | 33
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 |  |  | 4
  Not Hispanic or Latino | 4 | 2 | 15 | 3 | 7 | 2 | 0 | 13 |  |  | 46
  Missing | 1 | 1 | 4 | 1 | 5 | 1 | 3 | 3 |  |  | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White: White | 5 | 2 | 8 | 4 | 11 | 2 | 3 | 16 |  |  | 51
  White: Asian | 0 | 1 | 11 | 0 | 0 | 0 | 0 | 0 |  |  | 12
  White: Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 |  |  | 2
  White: Missing | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 |  |  | 4
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status has 3 Grades:
  0 - Asymptomatic (fully active, able to carry on all pre-disease activities without restriction)
  1. - Symptomatic but completely ambulatory (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  2. - Symptomatic, < 50% in bed during the day (ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours)
  Participants
    0 | 1 | 2 | 9 | 1 | 6 | 0 | 1 | 4 |  |  | 24
    1 | 3 | 1 | 9 | 1 | 4 | 2 | 2 | 10 |  |  | 32
    2 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 4 |  |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: DLT was defined as the occurrence of any of the following treatment-related toxicities, occurring through Day 28: Any grade ≥ 2 hemorrhagic event ; Any grade thrombocytopenia requiring PLT transfusion; PLT count < 25x109/L*; Grade 4 neutropenia (absolute neutrophil count < 0.5x109/L)*; Grade ≥ 3 febrile neutropenia*; Grade ≥ 2 total serum bilirubin with coincident direct bilirubin ≥ 0.5 mg/dL; Grade 3 non-hematologic toxicity for ≥ 7 consecutive days; Grade 4 non-hematologic toxicity. In the dose escalation stage in the core study period, the starting does in both strata was 5mg bid. Successive cohorts of newly enrolled patients received increasing doses of ruxolitinib until the Maximum Safe Starting Dose (MSSD) was determined. Initially, only patients with PLT counts 75-99 x10^9/L (stratum 1) were allowed to be enrolled. Once safety was established in stratum 1 at the first 2 dose cohorts, eligible population was further expanded to patients with PLT counts 50-74 x10^9/L (stratum 2).
Time Frame: 28 days
Population: Dose Determining Set. Dose was not escalated to enroll participants in Stratum-2 : Cohorts 4 and 5.
Measure: Count of Participants; unit: Participants
Groups:
- Stratum 1 : Cohort 1: Ruxolitinib was administered at 5 mg bid
- Stratum 1 : Cohort 2; Stratum 2 : Cohort 2: Ruxolitinib was administered at 5 mg q.AM+ 10 mg q.PM
- Stratum 1 : Cohort 3: Ruxolitinib was administered at a starting dose of 10 mg q.AM + 10 mg q.PM
- Stratum 1 : Cohort 4: Ruxolitinib was administered at a starting dose of 10 mg q.AM + 15 mg q.PM
- Stratum 1 : Cohort 5: Ruxolitinib was administered at a starting dose of 15 mg q.AM + 15 mg q.PM
- Stratum 2 : Cohort 1: Ruxolitinib was administered at 5 mg q.AM + 5 mg q.PM
- Stratum 2 : Cohort 3: Ruxolitinib was administered at 10 mg q.AM+ 10 mg q.PM
Arm/Group | Stratum 1 : Cohort 1 | Stratum 1 : Cohort 2 | Stratum 1 : Cohort 3 | Stratum 1 : Cohort 4 | Stratum 1 : Cohort 5 | Stratum 2 : Cohort 1 | Stratum 2 : Cohort 2 | Stratum 2 : Cohort 3
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 12 | 3 | 4 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAE's)
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Time Frame: approximately 4 years
Population: Full Analysis Population; Multiple dose cohorts within the strata are combined based on the total dose levels as specified in Statistical Analysis Plan
Measure: Count of Participants; unit: Participants
Groups:
- Stratum 1 : Group 1: Ruxolitinib was administered to Cohort 1 (5 mg bid) + Cohort 2 (5 mg q.AM / 10 mg q.PM) in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 1 : Group 2: Ruxolitinib was administered to cohort 3 at 10 mg bid in Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 1 : Group 3: Ruxolitinib was administered Cohort 4 (10 mg q.AM / 15 mg q.PM) + Cohort 5 (15 mg bid) in Participants with baseline Platelet counts of 75-99 x10^9/L.
- Stratum 2 : Group 1: Ruxolitinib was administered to Cohort 1 (5 mg bid) + Cohort 2 (5 mg q.AM / 10 mg q.PM) in participants with baseline Platelet counts of 50-74 x10^9/L
- Stratum 2 : Group 2: Ruxolitinib was administered Cohort 3 (10 mg bid) in participants with baseline Platelet counts of 50-74 x10^9/L
Arm/Group | Stratum 1 : Group 1 | Stratum 1 : Group 2 | Stratum 1 : Group 3 | Stratum 2 : Group 1 | Stratum 2 : Group 2
Number analyzed (Participants) | 8 | 20 | 16 | 7 | 18
Participants | 8 | 20 | 16 | 7 | 18

3. Secondary Outcome: Number of Subjects Achieving ≥ 50% Reduction in Palpable Spleen Length
Description: Participants achieving ≥ 50% reduction in palpable spleen length relative to study day 1 by treatment and stratum
Time Frame: 24 weeks
Population: All participants who had spleen assessment at week 24. Multiple dose cohorts within the strata are grouped according to total daily dose ranges as specified in Statistical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1 : Group 1 | Stratum 1 : Group 2 | Stratum 1 : Group 3 | Stratum 2 : Group 1 | Stratum 2 : Group 2
Number analyzed (Participants) | 5 | 15 | 13 | 5 | 8
Participants | 3 | 6 | 4 | 1 | 3

4. Secondary Outcome: Change in Spleen Length as Measure by Palpation Over Time
Description: Defined as measurement of change in spleen length by palpation from baseline
Time Frame: Day 8, 15, 22, 29, 43, 57, 85, 113, 141, 168, 252, 336, 420, 504, 588, 672, 756, 1008, 1092
Population: Change in spleen length measurement as compared to baseline are summarized by time and by stratum as specified in the SAP.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Stratum 1: Participants with baseline Platelet counts of 75-99 x10^9/L
- Stratum 2: Participants with baseline Platelet counts of 50-74 x10^9/L
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 44 | 25
cm
  Day 8: number analyzed (Participants) | 27 | 22
  Day 8 | -2.8 (2.73) | -3.7 (2.98)
  Day 15: number analyzed (Participants) | 42 | 25
  Day 15 | -3.3 (2.7) | -5.4 (4.4)
  Day 22: number analyzed (Participants) | 24 | 23
  Day 22 | -5.2 (2.87) | -5.4 (4.81)
  Day 29: number analyzed (Participants) | 43 | 25
  Day 29 | -4.4 (3.14) | -6.0 (4.23)
  Day 43: number analyzed (Participants) | 38 | 21
  Day 43 | -4.6 (2.74) | -5.8 (4.31)
  Day 57: number analyzed (Participants) | 39 | 22
  Day 57 | -4.5 (2.98) | -5.6 (4.52)
  Day 85: number analyzed (Participants) | 35 | 22
  Day 85 | -4.5 (3.53) | -5.2 (4.32)
  Day 113: number analyzed (Participants) | 34 | 22
  Day 113 | -4.7 (3.29) | -6.0 (4.74)
  Day 141: number analyzed (Participants) | 30 | 17
  Day 141 | -4.9 (3.24) | -6.7 (4.43)
  Day 168: number analyzed (Participants) | 33 | 13
  Day 168 | -5.2 (3.73) | -5.0 (4.78)
  Day 252: number analyzed (Participants) | 29 | 14
  Day 252 | -5.5 (4.40) | -3.6 (6.67)
  Day 336: number analyzed (Participants) | 22 | 14
  Day 336 | -5.1 (4.64) | -5.3 (4.86)
  Day 420: number analyzed (Participants) | 16 | 9
  Day 420 | -6.1 (4.80) | -4.9 (5.75)
  Day 504: number analyzed (Participants) | 20 | 8
  Day 504 | -5.7 (4.0) | -4.9 (4.91)
  Day 588: number analyzed (Participants) | 17 | 9
  Day 588 | -4.7 (5.24) | -5.4 (5.61)
  Day 672: number analyzed (Participants) | 18 | 9
  Day 672 | -5.8 (5.33) | -4.4 (6.60)
  Day 756: number analyzed (Participants) | 18 | 6
  Day 756 | -5.7 (5.22) | -6.0 (6.03)
  Day 1008: number analyzed (Participants) | 13 | 4
  Day 1008 | -7.6 (3.93) | -8.0 (4.55)
  Day 1092: number analyzed (Participants) | 4 | 5
  Day 1092 | -6.8 (1.71) | -4.2 (5.81)

5. Secondary Outcome: PK- C Reactive Protein Levels by PK Quartile (AUC0-12)
Description: To define the PK and C Reactive Protein relationship using PK Quartiles (AUC 0-12, ng*h/mL)
Time Frame: 24 weeks
Population: Results are summarized by strata, as dose relationship is accounted for by PK quartiles.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 44 | 25
micrograms/mL
  Quartile 1 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 1 Day 1 | 14 (5.73) | 12
  Quartile 1 Day 29: number analyzed (Participants) | 7 | 7
  Quartile 1 Day 29 | 21.2 (31.5) | 2.6 (2.05)
  Quartile 1 Day 168: number analyzed (Participants) | 4 | 7
  Quartile 1 Day 168 | 7.6 (8) | 5.51 (4.98)
  Quartile 2 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 2 Day 1 | 9.5 (0.707) | 7.7
  Quartile 2 Day 29: number analyzed (Participants) | 9 | 5
  Quartile 2 Day 29 | 10.2 (23.8) | 1.84 (173)
  Quartile 2 Day 168: number analyzed (Participants) | 7 | 4
  Quartile 2 Day 168 | 8.37 (12.8) | 2.41 (1.45)
  Quartile 3 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 3 Day 1 | 6.85 (7.28) | 6.5
  Quartile 3 Day 29: number analyzed (Participants) | 8 | 6
  Quartile 3 Day 29 | 2.76 (4.66) | 7.36 (9.06)
  Quartile 3 Day 168: number analyzed (Participants) | 6 | 5
  Quartile 3 Day 168 | 7.7 (14.9) | 4.98 (5.1)
  Quartile 4 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 4 Day 1 | 0.96 (1.05) | 5.4
  Quartile 4 Day 29: number analyzed (Participants) | 9 | 6
  Quartile 4 Day 29 | 1.87 (1.43) | 12.4 (17.8)
  Quartile 4 Day 168: number analyzed (Participants) | 11 | 1
  Quartile 4 Day 168 | 4.88 (9.01) | 4.9

6. Secondary Outcome: PK- Interleukin 1 Receptor Antagonist Levels by PK Quartile (AUC0-12)
Description: To define the PK and Interleukin 1 Receptor Antagonist relationship relationship using PK Quartiles (AUC 0-12, ng*h/mL)
Time Frame: 24 weeks
Population: Results are summarized by strata, as dose relationship is accounted for by PK quartiles.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 44 | 25
picograms/mL
  Quartile 1 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 1 Day 1 | 188 (116) | 105
  Quartile 1 Day 29: number analyzed (Participants) | 7 | 7
  Quartile 1 Day 29 | 267 (334) | 588 (730)
  Quartile 1 Day 168: number analyzed (Participants) | 4 | 7
  Quartile 1 Day 168 | 592 (532) | 379 (419)
  Quartile 2 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 2 Day 1 | 179 (43.1) | 133
  Quartile 2 Day 29: number analyzed (Participants) | 9 | 5
  Quartile 2 Day 29 | 524 (519) | 600 (649)
  Quartile 2 Day 168: number analyzed (Participants) | 7 | 4
  Quartile 2 Day 168 | 557 (504) | 334 (322)
  Quartile 3 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 3 Day 1 | 319 (288) | 191
  Quartile 3 Day 29: number analyzed (Participants) | 8 | 6
  Quartile 3 Day 29 | 304 (327) | 452 (529)
  Quartile 3 Day 168: number analyzed (Participants) | 6 | 5
  Quartile 3 Day 168 | 549 (531) | 960 (792)
  Quartile 4 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 4 Day 1 | 120 (40.3) | 148
  Quartile 4 Day 29: number analyzed (Participants) | 9 | 6
  Quartile 4 Day 29 | 604 (647) | 475 (464)
  Quartile 4 Day 168: number analyzed (Participants) | 11 | 1
  Quartile 4 Day 168 | 562 (758) | 378

7. Secondary Outcome: PK- Tissue Necrosis Factor Receptor 2 Levels by PK Quartile (AUC0-12)
Description: To define the PK and Tissue Necrosis Factor Receptor 2 relationship using PK Quartiles (AUC 0-12, ng*h/mL)
Time Frame: 24 weeks
Population: Results are summarized by strata, as dose relationship is accounted for by PK quartiles.
Measure: Mean (Standard Deviation); unit: nanograms/mL
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 44 | 25
nanograms/mL
  Quartile 1 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 1 Day 1 | 24 (19.8) | 6.2
  Quartile 1 Day 29: number analyzed (Participants) | 7 | 7
  Quartile 1 Day 29 | 20.5 (19.7) | 25.7 (14.4)
  Quartile 1 Day 168: number analyzed (Participants) | 4 | 7
  Quartile 1 Day 168 | 14 (4.24) | 22.6 (12.6)
  Quartile 2 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 2 Day 1 | 13.5 (0.707) | 8.2
  Quartile 2 Day 29: number analyzed (Participants) | 9 | 5
  Quartile 2 Day 29 | 14.9 (6.62) | 12.3 (7.67)
  Quartile 2 Day 168: number analyzed (Participants) | 7 | 4
  Quartile 2 Day 168 | 36.1 (22.9) | 18.4 (12.6)
  Quartile 3 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 3 Day 1 | 21 (9.9) | 47
  Quartile 3 Day 29: number analyzed (Participants) | 8 | 6
  Quartile 3 Day 29 | 12.9 (4.32) | 13.7 (11.6)
  Quartile 3 Day 168: number analyzed (Participants) | 6 | 5
  Quartile 3 Day 168 | 13.3 (5.8) | 12.4 (7.99)
  Quartile 4 Day 1: number analyzed (Participants) | 2 | 1
  Quartile 4 Day 1 | 15 (4.24) | 24
  Quartile 4 Day 29: number analyzed (Participants) | 9 | 6
  Quartile 4 Day 29 | 15.7 (9.13) | 24.6 (17.4)
  Quartile 4 Day 168: number analyzed (Participants) | 11 | 1
  Quartile 4 Day 168 | 14.3 (7.67) | 11

8. Secondary Outcome: AUC 0-Inf
Description: Area Under the Serum Concentration Versus Time Curve，Time 0 to Infinity
Time Frame: 0.25 to 0.75, 1 to 3, and 4 to 12 hours postdose on Day 1 and predose, 0.25 to 0.75 hours, and 1 to 3 hours postdose on Day 15, with a random sample on Days 29 and 57
Population: Results are summarized by strata; dose relationship is accounted for by PK quartile grouping.
Measure: Mean (Standard Deviation); unit: nM*hr
Groups:
- 5mg BID: ruxolitinib was administered at 5 mg BID
- 10mg BID: ruxolitinib was administered at 10 mg BID
- 15 mg BID: ruxolitinib was administered at 15 mg BID
Arm/Group | 5mg BID | 10mg BID | 15 mg BID
Number analyzed (Participants) | 15 | 16 | 9
nM*hr | 1027 (357) | 1930 (562) | 3756 (916)

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: AE additional description
Arm/Group | Stratum 1 : Cohort 1 | Stratum 1 : Cohort 2 | Stratum 1 : Cohort 3 | Stratum 1 : Cohort 4 | Stratum 1 : Cohort 5 | Stratum 2 : Cohort 1 | Stratum 2 : Cohort 2 | Stratum 2 : Cohort 3 | Stratum 2 : Cohort 4 | Stratum 2 : Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 3/20 | 1/4 | 0/12 | 1/3 | 0/4 | 4/18 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/3 | 10/20 | 4/4 | 5/12 | 3/3 | 3/4 | 9/18 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 20/20 | 4/4 | 12/12 | 3/3 | 4/4 | 18/18 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stratum 1 : Cohort 1 (N=5) | Stratum 1 : Cohort 2 (N=3) | Stratum 1 : Cohort 3 (N=20) | Stratum 1 : Cohort 4 (N=4) | Stratum 1 : Cohort 5 (N=12) | Stratum 2 : Cohort 1 (N=3) | Stratum 2 : Cohort 2 (N=4) | Stratum 2 : Cohort 3 (N=18) | Stratum 2 : Cohort 4 (N=0) | Stratum 2 : Cohort 5 (N=0)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0/0 | 0/0 | 0/0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 2 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Stratum 1 : Cohort 1 (N=5) | Stratum 1 : Cohort 2 (N=3) | Stratum 1 : Cohort 3 (N=20) | Stratum 1 : Cohort 4 (N=4) | Stratum 1 : Cohort 5 (N=12) | Stratum 2 : Cohort 1 (N=3) | Stratum 2 : Cohort 2 (N=4) | Stratum 2 : Cohort 3 (N=18) | Stratum 2 : Cohort 4 (N=0) | Stratum 2 : Cohort 5 (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 11 | 2 | 6 | 1 | 3 | 8 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 9 | 3 | 11 | 1 | 4 | 14 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 2 | 1 | 0 | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 6 | 2 | 3 | 1 | 2 | 5 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0/0 | 0/0 | 0/0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 3 | 0 | 2 | 2 | 0 | 5 | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Fatigue (General disorders) | 0 | 0 | 3 | 1 | 3 | 0 | 1 | 3 | NA | NA
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Influenza like illness (General disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | NA | NA
Oedema peripheral (General disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 3 | NA | NA
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA
Pyrexia (General disorders) | 1 | 0 | 6 | 0 | 2 | 2 | 1 | 4 | NA | NA
Swelling face (General disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | NA | NA
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Herpes virus infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | NA | NA
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 1 | 4 | 1 | 1 | 0 | 1 | 5 | NA | NA
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0/0 | 0/0 | 0/0 | NA | NA
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | NA | NA
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 2 | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | NA | NA
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 2 | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | NA | NA
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0/0 | 0/0 | 0/0 | NA | NA
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Coagulation factor V level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Coagulation factor VII level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Coagulation factor X level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | NA | NA
Haemoglobin decreased (Investigations) | 0 | 0 | 4 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Platelet count decreased (Investigations) | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 1 | NA | NA
Prothrombin level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Prothrombin time shortened (Investigations) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Red blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Weight increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | NA | NA
White blood cell count decreased (Investigations) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 2 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 5 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 2 | 1 | 3 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 3 | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | NA | NA
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 3 | 1 | 1 | 4 | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | NA | NA
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0/0 | 0/0 | 0/0 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 3 | 2 | 2 | 6 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5 | 1 | 2 | 0 | 1 | 0 | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 6 | 0 | 0 | 1 | 1 | 2 | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 1 | NA | NA
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | NA | NA
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | NA | NA
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0/0 | 0/0 | 0/0 | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 3 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | 0 | 0
Platelet aggregation inhibition (Blood and lymphatic system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | NA | NA
Malaise (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | NA | NA
Mucosal inflammation (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Oedema (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | NA | NA
Xerosis (General disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Jaundice (Hepatobiliary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Campylobacter infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Cystitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Escherichia urinary tract infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Folliculitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Herpes simplex (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Herpes zoster (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Influenza (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 2 | NA | NA
Oropharyngeal candidiasis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | NA | NA
Periodontitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Pharyngitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Pharyngotonsillitis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Vulvovaginal candidiasis (Infections and infestations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Anaemia postoperative (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Ligament sprain (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | NA | NA
Scratch (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 0 | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Tooth fracture (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Wound (Injury, poisoning and procedural complications) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Amylase increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Blood calcium decreased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Blood urea increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Cardiac murmur (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Lipase increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Urine output increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
White blood cell count increased (Investigations) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Gout (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Iron overload (Metabolism and nutrition disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 2 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Memory impairment (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 2 | NA | NA
Presyncope (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Somnolence (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Tremor (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | NA | NA
Depression (Psychiatric disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 2 | NA | NA
Dysuria (Renal and urinary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Haematuria (Renal and urinary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Erectile dysfunction (Reproductive system and breast disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 1 | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 1 | NA | NA
Rales (Respiratory, thoracic and mediastinal disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Pain of skin (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Skin discolouration (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Haemorrhage (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Hot flush (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA
Pallor (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 2 | NA | NA
Peripheral ischaemia (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 1 | 0 | NA | NA
Systolic hypertension (Vascular disorders) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0 | 0 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT01317875/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT01317875/SAP_001.pdf